CLINICAL TRIAL: NCT03524183
Title: The Virtual Fitness Buddy Ecosystem: Using Digital Technology to Promote and Sustain Moderate-to-Vigorous Intensity Physical Activity in Children
Brief Title: Virtual Fitness Buddy Ecosystem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: YMCA of Metropolitan Atlanta (Other)
Responsible Party: Principal Investigator, Sun Joo (Grace) Ahn, PHD, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00004611
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The efficacy of the VFB Ecosystem will be tested using a cluster randomized trial with repeated measures at baseline, posttest (immediately after 3-month intervention), mid-term follow up (6 months post intervention), and a long-term follow up (12 months post intervention). A 3-month intervention period was selected to observe variance in engagement over the course of an academic semester in the afterschool programs. A cluster randomized design is indicated when outcomes are tracked at a group level (afterschool programs) instead of at the individual level (children) and is the preferred method to reduce the impact of dependency in the data. From a pool of 24 demographically matched afterschool programs, we will randomly assign pairs to either receive the Ecosystem or physical activity as usual. Outcomes will be modeled and expressed as changes occurring at the afterschool program level--the unit of randomization.
Who Masked: Participant
Masking Description: The unit of randomization (control vs. treatment) is at the school level. Participants at each school will be masked of the other schools' assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The children will receive the standard of care at their respective afterschool programs. As with the treatment group, all children will be asked to wear their Fitbits for one year following the intervention period, for the mid- and long-term follow up. Fitbit data will be recorded tracked year-round through the automated Fitbit data syncing stations at the afterschool program site. All participants will be assessed for PA and psychosocial variables at the same four measurement points for the treatment group.
  Interventions: Behavioral: Virtual Fitness Buddy Ecosystem
- Treatment (Experimental): The virtual pet functions as a personalized fitness buddy to encourage children to set and meet physical activity goals, promote physical activity self-efficacy, and foster mutually supportive relationships among children, parents, and the virtual pet. Concurrently, the kiosk sends a text message to parents on the child's physical activity progress. Parents are then able to send words of encouragement and communicate with their children via the kiosk, using the text messaging feature of their mobile phones. Parents will also receive text messages from the kiosk with a security code to access a website that provides detailed records of the child's physical activity over time. Participants will be assessed for post-treatment measurements immediately after 3 months, 6 months after, and 12 months after the intervention.
  Interventions: Behavioral: Virtual Fitness Buddy Ecosystem

INTERVENTIONS:
Behavioral: Virtual Fitness Buddy Ecosystem — The Virtual Fitness Buddy Ecosystem allows parents to stay involved in the intervention and support their children's PA efforts even when they cannot be with their children. A virtual pet, designed to mimic human-pet relationships in the physical world, will guide children to set and meet PA goals and offer tailored support. In collaboration with YMCA, 480 children and 480 parents in 24 afterschool programs will be randomly assigned to treatment and control groups. Afterschool programs in the treatment group will receive the Ecosystem intervention for 6-months; afterschool programs in the control group will not experience the Ecosystem. All children will complete baseline assessments, a 3-month posttest, and a 6-month and 12-month follow up. Parents and children will provide self-report data on their perceived social support, motivation, and PA self-efficacy. PA will be assessed with activity monitors, which children will wear throughout the project.

SUMMARY:
The VFB Ecosystem capitalizes on digital technologies' ability to connect parents and children, allowing parents to actively support their child's physical activity, even when parents cannot be present. The VFB is a kiosk-based system that houses a virtual dog programmed to allow children to set self-determined physical activity goals. The children wear Fitbits while performing physical activity. Using the unique data embedded in the Fitbit, the kiosk is able to detect each individual child and automatically connect him or her to a unique, personalized virtual dog. Physical activity data is transmitted automatically from the Fitbit to the kiosk when the child approaches, and the virtual dog provides accurate evaluations of whether the child met the self-determined physical activity goal, offering words of encouragement and physical activity support. The virtual pet functions as a personalized fitness buddy to encourage children to set and meet physical activity goals, promote physical activity self-efficacy, and foster mutually supportive relationships among children, parents, and the virtual pet. This will be particularly helpful for children who receive insufficient amounts of social support in their current environment.

Concurrently, the kiosk sends a text message to parents on the child's physical activity progress. Parents are then able to send words of encouragement and communicate with their children via the kiosk, using the text messaging feature of their mobile phones. Thus, even when the parent is not with the child, the virtual pet is designed to serve as a coordinating focus for facilitating parent-child communication. Parents will also receive text messages from the kiosk with a security code to access a website that provides detailed records of the child's physical activity over time.

DETAILED DESCRIPTION:
Childhood obesity poses a critical public health concern and chronically remains as one of the strongest predictors of obesity as an adult. Scientific evidence has demonstrated that daily physical activity (PA) is imperative in preventing the onset of obesity. The outpour of academic and professional interest has increased the public awareness of the risks related to obesity (e.g., type 2 diabetes, cardiovascular diseases, cancers) as well as the importance of PA. However, studies show that the rising prevalence of childhood obesity has not faltered since 1999. Many existing PA interventions show short-term impact, but have failed to demonstrate longer-term efficacy in sustaining the changes in PA over time-a gap this project aims to address.

One important, yet commonly overlooked, limitation of existing PA interventions is the negative impact of extrinsic rewards, such as points, grades, and badges, which are often used in health promotion interventions to incentivize children for engaging with the program. Children become motivated to excel in obtaining the extrinsic rewards rather than learning the intrinsic benefits of the intervention. Consequently, these types of interventions have limited effects that may disappear altogether when they stop receiving extrinsic rewards. Another critical limitation of existing PA interventions related to the use of extrinsic rewards is that the focus on "beating the system" by obtaining extrinsic rewards decontextualizes the intervention from the child's everyday life. This is an isolating experience for the child, taking him or her away from existing social support (e.g., parents) and left to his or her devices to engage in PA, based solely on the motivation from extrinsic rewards.

Guided by the frameworks of social ecological theory and self-determination theory, we propose a paradigm-shifting intervention through an engaging, game-like platform that incorporates intrinsic reward systems by harnessing the power of technology to connect people and devices to promote PA in children. The Virtual Fitness Buddy (VFB) Ecosystem was designed to encourage children to embrace PA as a lifestyle change that can be sustained over time rather than a means to gain points. The Ecosystem meets this goal by leveraging one of the most influential existing social relationships in children's lives, the parent-child relationship. Using consumer-grade technological devices, such as mobile phones, the Ecosystem allows parents to stay involved in the intervention and support their children's PA efforts even when they cannot be with their children. In addition, a virtual pet, designed to mimic human-pet relationships in the physical world, will guide children to set and meet PA goals and offer tailored support.

Using technology to amplify the power of existing social relationships, children will learn to embrace PA as a lifestyle change while supported by their parents and the virtual pet within the Ecosystem. Because the intervention is embedded in the context of children's everyday lives, our preliminary findings demonstrated the potential of the Ecosystem to elicit high levels of engagement and excitement from both children and parents over a 3-day intervention period. The next critical question is whether the Ecosystem can maintain children and parents' engagement over longer periods of time, yielding sustainable changes in health behavior and lifestyle choices that were initiated by the Ecosystem.

In collaboration with YMCA, 480 children and 480 parents in 24 afterschool programs will be randomly assigned to treatment and control groups in a cluster-randomized controlled trial. Afterschool programs in the treatment group will receive the Ecosystem intervention for 3-months; afterschool programs in the control group will not experience the Ecosystem (but will receive the standard of care). All children will complete baseline assessments, a 3-month posttest, and a 6-month and 12-month follow up. Parents and children will provide self-report data on their perceived social support, motivation, and PA self-efficacy. PA will be assessed with activity monitors, which children will wear throughout the project.

Our specific aims are:

Aim 1. Test the hypothesis that at the 3-month, 6 month, and 12-month assessments, children assigned to the Ecosystem will evince higher levels of moderate-to-vigorous intensity PA than children in the control group.

Auxiliary Aim 1. For the treatment group only, test the engagement of parents and children over the 3-month intervention through tracking the usage frequency and duration of their interactions through the Ecosystem.

Aim 2. Test the parent and child mechanisms of change. Specifically, we hypothesize that children and parents in the treatment group will report higher levels of motivation, PA self-efficacy, and perceived social support at the 3-month, 6 month, and 12-month follow up compared to control children. Moderators of change, such as the child's age and gender will also be analyzed.

The Virtual Fitness Buddy Ecosystem represents a new generation of technology-mediated health interventions for children, which integrates fun and engaging technology into existing social systems, to promote sustainable lifestyle changes through the intrinsic reward of social support. Because the Ecosystem is a cost- and labor-effective solution that integrates consumer-grade technology with low barriers for continued use, it has the potential for rapid diffusion and widespread public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between the ages of 6-10
* Children must be daily participants in the specified afterschool program
* Only one child (oldest) and one caregiver from each family can participate
* Participating parent must be the caregiver for the child for the majority of the week

Exclusion Criteria:

* Family has imminent plans for moving
* Child has impairments that prevent unassisted physical activity
* A non-residential parent who has little interaction with the child

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 964 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 12 months
  Physical activity of participating children will be assessed with Fitbits and validated with Actigraphs.
Height | 12 months
  Height in meters
Weight | 12 months
  Weight in kilograms
Waist circumference | 12 months
  Waist circumference in centimeters
Body fat percentage | 12 months
  Body fat percentage in percentile
Self-efficacy | 12 months
  Self-reported perceived efficacy for physical activity
Motivation | 12 months
  Self-reported motivation for physical activity
Parent-child relationship | 12 months
  Self-reported parent-child relationship

CONTACTS AND LOCATIONS:
Overall Officials: Sun Joo (Grace) Ahn, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- YMCA of Metropolitan Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The overriding aim of this project is to help tackle the childhood obesity epidemic, which of national importance. As such, all of the investigators are committed to ensuring widespread dissemination of our findings and to making the technologies developed freely available to other researchers. This will include publishing not just our evaluation results through appropriate scholarly journals and presentations at national meetings, but also our experiences and lessons learned during the design and development process. For example, our design documents will evolve on password-protected website that, upon completion of the project, will be made public (with teacher names removed) with contact details for the investigators included, and will be detailed in publications and presentations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Data files will be compiled as data collection progresses. After completion of the study, data analysis, and manuscript publication, the PI will share de-identified data with researchers who can verify certification to (a) work with Human Subjects and (b) complete an agreement with the host institution, the University of Georgia. Thus, following study completion, all data will be accessible to qualified researchers. Additionally, surveys created for the study will be hosted on university websites to be used free of charge by interested researchers. Treatment manuals and other materials will be made available upon request.